CLINICAL TRIAL: NCT00023049
Title: Genetic Analysis of Hereditary Disorders of Hearing and Balance
Status: Completed | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010229; 01-DC-0229
Record Dates: First submitted 2001-08-21; First posted 2001-08-22 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-02-26

CONDITIONS: Sensorineural Hearing Loss; Hearing Disorder; Vestibular Disease
Keywords: Deafness; Phenotypes; Natural History Study; Auditory; DNA Mutations; Natural History; Hereditary Hearing Disorder; Hearing Impairment; Sensorineural Hearing Loss; Vestibular Dysfunction; SNHL
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Disorders; Vestibular Diseases; Deafness; Hearing Loss

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patients with known SNHL and/or peripheral vestibular dysfunction

SUMMARY:
This study will try to identify the genetic causes of hereditary hearing loss or balance disorders.

People with a hearing or balance disorder that affects more than one family member may be eligible for this study. They and their immediate family members may undergo some or all of the following procedures:

* Medical and family history, including questions about hearing, balance and other ear-related issues, and review of medical records.
* Routine physical examination.
* Blood draw or buccal swab (brushing inside the cheek to collect cells) - Tissue is collected for DNA analysis to look for changes in genes that may be related to hearing loss.
* Hearing tests - The subject listens for tones emitted through a small earphone.
* Balance tests to see if balance functions of the inner ear are associated with the hearing loss In one test the subject wears goggles and watches moving lights while cold or warm air is blown into the ears. A second test involves sitting in a spinning chair in a quiet, dark room.
* Photograph - A photograph may be taken as a record of eye shape and color, distance between the eyes, and hair color.
* Computed tomography (CT) and magnetic resonance imaging (MRI) scans - These tests show the structure of the inner ear. For CT, the subject lies still for a short time while X-ray images are obtained. For MRI, the patient lies on a stretcher that is moved into a cylindrical machine with a strong magnetic field. The magnetic field and radio waves produce images of the inner ear. The radio waves cause loud thumping noises that can be muffled by the use of earplugs.

DETAILED DESCRIPTION:
Hereditary hearing impairment is a genetically heterogeneous disorder that can be caused by mutations in any one of hundreds of different genes. Approximately 120 genes have now been identified in which mutations can cause nonsyndromic sensorineural hearing loss. The identification and analysis of these genes and their mutations are providing critical insights into the development, structure, and function of the auditory system, as well as the molecular mechanisms associated with disruption of these processes. In contrast, the molecular mechanisms underlying familial disorders affecting peripheral vestibular function appear to be more rare, have not been well described, and are less well understood. The peripheral auditory and vestibular systems share many common features in both health and disease, and many hereditary hearing loss disorders also affect vestibular function. The purpose of this study is to identify genes and mutations causing hereditary disorders of hearing, balance, or both. Members of families segregating hereditary disorders of hearing or balance will be enrolled in the proposed study in order to: (1) define and characterize the phenotypes and natural histories; (2) identify the underlying causative mutations and genes by linkage, positional cloning, and/or candidate gene mutation analyses; (3) and correlate observed phenotypes with the corresponding mutations and functions of the underlying genes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Persons with known SNHL and/or peripheral vestibular dysfunctions caused by genetic etiology

Family members of persons with known SNHL and/or peripheral vestibular dysfunction caused by genetic etiology

Adults must be able to provide informed consent

Minors must have a parent or guardian able to provide informed consent

Subjects must be 0-99 years of age

For Nigeria subjects with non-syndromic hearing loss, their hearing loss must be early-onset, before 10 years of age, to be eligible.

EXCLUSION CRITERIA:

Persons with SNHL and/or peripheral vestibular dysfunction caused by a nongenetic etiology such as trauma, infection, metabolic or immunologic disorders, or exposure to ototoxic agents such as noise or aminoglycoside antibiotics will not be included in this protocol.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will be studying up to 750 people with hearing losses or balance problems that are thought to be hereditary and, if possible, their family members, either with or without hearing or balance problems to participate in our study. A total of up to 400 affected and unaffected individuals, including family members and control subjects will be enrolled from the Nigerian population.
Sampling Method: Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2002-12-23 (Actual)

PRIMARY OUTCOMES:
To define and characterize the phenotypes and natural histories of families with segregating hereditary disorders of balance or hearing and to identify the possible mutations and genes by genetic analysis | Ongoing
  Characterize the natural history of hereditary disorders affecting hearing and/or balance Identify the genes, including both known and as yet undiscovered genes, that can cause hereditary disorders of hearing or balance Identify and characterize the structure and functions of these genes in the development and function of the peripheral auditory and vestibular systems Determine how mutations in these genes cause hearing loss and vestibular dysfunction Correlate genotypes and phenotypes to identify clinical features that may be used to facilitate the genetic diagnosis of hereditary disorders affecting hearing or balance

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Friedman, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (2):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Institute of Child Health, College of Medicine, University of Ibadan, Ibadan, Nigeria

REFERENCES:
- [Background] Cohn ES, Kelley PM, Fowler TW, Gorga MP, Lefkowitz DM, Kuehn HJ, Schaefer GB, Gobar LS, Hahn FJ, Harris DJ, Kimberling WJ. Clinical studies of families with hearing loss attributable to mutations in the connexin 26 gene (GJB2/DFNB1). Pediatrics. 1999 Mar;103(3):546-50. doi: 10.1542/peds.103.3.546. PMID 10049954
- [Background] Griffith AJ, Friedman TB. Making sense out of sound. Nat Genet. 1999 Apr;21(4):347-9. doi: 10.1038/7668. No abstract available. PMID 10192378
- [Background] Morton NE. Genetic epidemiology of hearing impairment. Ann N Y Acad Sci. 1991;630:16-31. doi: 10.1111/j.1749-6632.1991.tb19572.x. No abstract available. PMID 1952587
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-DC-0229.html